CLINICAL TRIAL: NCT06519656
Title: A Clinical Efficacy Study of Mazdutide in the Treatment of Polycystic Ovary Syndrome
Brief Title: Efficacy of Mazdutide for Treating PCOS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-190R2
Record Dates: First submitted 2024-07-14; First posted 2024-07-25 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — mazdutide; Glucagon-Like Peptide-1 Receptor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mazdutide Treatment Arm (Experimental): Subcutaneous injection of Mazdutide once weekly for 24 weeks.
  Interventions: Drug: Mazdutide

INTERVENTIONS:
Drug: Mazdutide — In the initial 4 weeks, the subjects are given Mazdutide 2mg once weekly. If well tolerated, the dosage is increased to 4mg once weekly for another 4 weeks. If still well tolerated, the dosage is further increased to 6mg once weekly and maintained for the ensuing 16 weeks.
  Other Names: GLP-1R and GCGR dual agonist

SUMMARY:
The goal of this clinical trial is to learn the efficacy of Mazdutide in treating obese female adults diagnosed with polycystic ovary syndrome (PCOS). The main question it aims to answer is: Does Mazdutide lower the free androgen index (FAI) in obese female adults with PCOS? Participants will take Mazdutide once every week for 24 weeks and visit the clinic once every 4 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥28kg/M2
* No plan for pregnancy in the coming 8 months after enrollment
* Patients should meet at least two of the three criteria according to the 2023 international evidence-based guideline for PCOS :

  1. Irregular cycles and ovulatory dysfunction: < 21 or > 35 days or < 8 cycles per year; > 90 days for any one cycle
  2. Polycystic ovaries: ≥20 follicles in at least one of two ovaries (diameter<10mm), confirmed by ultrasound
  3. Biochemical hyperandrogenism: total testosterone>1.67 nmol/L or clinical hyperandrogenism: modified Ferriman Gallwey score (mFG)>4

Exclusion Criteria:

* Previous history of acute or chronic pancreatitis or pancreatic injury
* Previous history or family history of medullary thyroid cancer, multiple endocrine neoplasia type 2a or 2b
* Severe hypertriglyceridemia (TG>5mmol/L)
* Type 1 or type 2 diabetes mellitus
* Other endocrine diseases that can cause secondary PCOS, including but not limited to: 21 hydroxylase deficiency, prolactinoma, hypothyroidism, Cushing's syndrome, etc
* Pregnancy or breast-feeding
* Patients with other serious diseases affecting heart, liver, kidney, or other major organs
* Patients with any type of cancer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Free Androgen Index (FAI) | 24 weeks
  FAI=total testosterone (nmol/L)/ sex hormone binding globulin (nmol/L) X 100

SECONDARY OUTCOMES:
Times of regular menses | 24 weeks
  Record of vaginal bleeding within 24 weeks after using Mazdutide
Number of immature follicles | 24 weeks
  Total number of follicles measuring 2-9 mm in diameter on ultrasound
Bilateral ovary volume | 24 weeks
  Total ovary volume is calculated based on length, width and height of bilateral ovaries measured by ultrasound
Serum anti-Mullerian hormone (AMH) | 24 weeks
  Measurement of serum AMH
HOMA insulin resistance index (HOMA-IR) | 24 weeks
  HOMA-IR=fasting plasma glucose (mmol/L)×fasting insulin (μU/mlINS)/22.5
HbA1c | 24 weeks
  Measurement of HbA1c
body mass index (BMI) | 24 weeks
  BMI = weight / height² (weight in kilograms and height in meters)

CONTACTS AND LOCATIONS:
Overall Officials: XI DONG, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No